CLINICAL TRIAL: NCT04252170
Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly (Feasibility Study)
Brief Title: Arm Motor Rehabilitation, Entertainment and Cognition System for the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bright Cloud International Corp (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Genesis HealthCare System (Other)
Responsible Party: Principal Investigator, Dr. Nam H. Kim, Director of Engineering, Bright Cloud International Corp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BCI-10-001; 5R44AG044639-05 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Rehabilitation

STUDY DESIGN:
Intervention Model Description: 6 will be stroke survivors inpatients at PowerBack, Piscataway NJ, USA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Feasibility study, Stroke Survivors (Experimental): BAC feasibility study at PowerBack, Piscataway NJ, with stroke patients.
  Interventions: Device: Rehabilitation Therapy, Experimental on the BrightArm Compact device

INTERVENTIONS:
Device: Rehabilitation Therapy, Experimental on the BrightArm Compact device — Experimental group will receive VR game-based rehabilitation therapy through Bright Cloud's proprietary device, called BrightArm Compact (BAC). An Occupational Therapist will assist as needed.
  Other Names: BrightArm Compact rehabilitation through games

SUMMARY:
The research project is intended to provide information pertaining to the feasibility of the BrightArm Compact robotic rehabilitation system for patients early sub-acute post Cerebral Vascular Accident. The aims are to: a) determine clinical benefit to motor and cognitive function as well as mood; 2) to ascertain technology acceptance by patients and therapists. The experimental training consists of 12 integrative arm/hand and cognitive training by playing therapeutic games. Participants are evaluated pre-and post-intervention and provide subjective evaluation of the system.

DETAILED DESCRIPTION:
This study targets participants, who had suffered a first stroke recently, and who may or may not have been diagnosed with mild cognitive impairments or dementia (including Alzheimer's disease). It is important to find out if these improvements can be obtained with the computer game-based integrative (motor-cognitive) bilateral rehabilitation developed by Bright Cloud International Corp, and if these gains transfer to daily activities.

Specific aims are:

* BAC technology acceptance;
* improvement in motor function for the upper extremity;
* strengthening of shoulder and fingers;
* increased active (self initiated) range of motion for shoulder, arms and fingers;
* improved independence in activities of daily living;
* improvement in cognitive areas of memory, attention and decision making;
* improved mood (as in reduced depression severity);

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 85;
* diagnosis of first-time CVA that occurred more than 5 days prior and less than 21 days prior
* English speakers;
* UE unilateral or bilateral involvement (from new bilateral CVA)
* motor involvement (FMA score 20 to 45);
* ability to actively move UE more than 10 degrees for shoulder and elbow flexion/extension;
* ability to actively extend fingers at least 5 degrees
* cognitive skills to participate (Montreal Cognitive Assessment (MoCA) [Nasreddine et al 2005] score 10-30).
* Subjects may have normal cognition, MCI or dementia

Exclusion Criteria:

* being younger than 50 or older than 85 years of age
* previous stroke
* Stroke that occurred more than 20 days prior to enrollment
* Inability to actively extend fingers at least 5 degrees;
* Fugl-Meyer scores of 19 or less;
* severe visual neglect or legally blind
* severe hearing loss or deafness
* receptive aphasia or severe expressive aphasia;
* severe spasticity (Modified Ashworth Scale 4/4)
* contractures of the upper limb joints
* uncontrolled hypertension (>190/100 mmHg)
* severe cognitive impairment determined by Montreal Cognitive Assessment (MoCA) [Nasreddine et al, 2005] test of 9 and below;
* No chemodenervation or nerve block to upper limb involved during the experimental period (e.g., botulinum toxin injection)
* inability to speak English;
* a history of violence or drug abuse;
* paranoia and psychotic behavior;
* inability participate in the neuropsychological pre-study assessment for reliable scores (e.g., cognitive impairment, communication disorders).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Artificial Intelligence-determined game difficulty level | Through study completion, an average of 3 weeks
  BrightBrainer game difficulty setting is determined based on patient's past performance, in order to adapt the therapy to a given individual. It representing an average or difficulties of all games played in a session. The measure implies game play intensity and level of challenge
Game Score (baseline and performance) | Through study completion, an average of 3 weeks
  BrightBrainer game baseline and performance scores. Min. score is 0. Max depends on specific game.
Participants' feedback using 5-point Likert scale | Through study completion, an average of 3 weeks
  Subjective evaluation feedback and overall ratings on BrightBrainer games. Consists of multiple questions, each ranked on a 5-point Likert scale, with 1 (min) and 5 (max).
Therapist subjective evaluation using 5-point Likert scale | 3 weeks
  Subjective evaluation given by the attending Occupational Therapist at the end of the experimental intervention. Multiple questions, each ranked from 1 (min) to 5 (max)

SECONDARY OUTCOMES:
Arm Range of Motion | Change from Baseline arm range of motion at 3 weeks
  measurement of active movement initiated by participant using a mechanical goniometer
Finger Range of Motion | Change from Baseline finger range of motion at 3 weeks
  finger extension/flexion range using a mechanical goniomter
Grasp Strength with Jamar Dynamo-meter | Change from Baseline grasp strength at 3 weeks
  grasp strength measurement using dynamo-meter
Pinch strength with pinch meter | Change from Baseline at 3 weeks
  Pinch strength measured with fingers placed on a pinch meter
Shoulder strength | Change from Baseline shoulder strength at 3 weeks
  Measurement of shoulder strength using calibrated wrist weights
Fugl-Meyer Assessment (Upper Extremity sub-scale) score | Change from Baseline Fugl-Meyer Assessment Score at 3 weeks
  Upper Extremity Motor function, score scale is 0 (min) to 66 (max). Larger score means better outcome.
Upper extremity functional index (UEFI) score | Change from Baseline Upper Extremity Functional Inex score at 3 weeks
  A self report of independence in 20 activities of daily living (ADLs). Total score range is 0 (min) to 80 (max). Larger score means better outcome.
CAHAI 9 Score | Change from Baseline CAHAI 9 score at 3 weeks
  Chedoke Arm and Hand Activity Inventory, reflecting ADL independence in simulated bimanual activities. Min score 9, max score 63, with larger score meaning better outcomes.
Jebsen Test of Hand Function | Change from Baseline Jebsen Test of Hand Function score at 3 weeks
  Timed test of 7 simulated activities of daily living. Lowest score is 0, largest score is 1260. Units are seconds. Lower score means better outcomes (faster completion).
Beck Depression Inventory II (BDI II) score | Change from Baseline depression severity at 3 weeks
  participants' depression measure. Range is 0 (min) to 63 (max). Lower score indicate better outcomes (less depression).
Verbal attention | Change from Baseline verbal attention at 3 weeks
  Attention module digit span (working memory) in the Neuropsychological Assessment Battery NAB min 0, larger score is better
Verbal fluency | Change from Baseline verbal fluency at 3 weeks
  verbal fluency test min 0, larger score is better
Verbal memory | Change from Baseline verbal learning memory at 3 weeks
  Hopkins Verbal Learning Test, Revised (HVLT-R) min 0, larger is better
Brief Visuospatial Memory Test-Revised | Change from Baseline visuospatial memory at 3 weeks
  A measure of memory function min 50 std of 10, larger score is better
Executive Function Module | Change from Baseline executive function at 3 weeks
  Word Generation min 0, larger is better
Cognitive executive function | Change from Baseline Trail Making Test B (TMT-B) Score at 3 weeks
  Trail Making Test B (TMT-B) lMin 50, std of 10, larger number means better outcomes
Cognitive executive function | Change from Baseline NAB Exec Score at 3 weeks
  NAB Executive Functioning Module min 50, std is 10, larger number means better outcomes
Visual attention | Change from Baseline visual attention at 3 weeks
  Attention module dots (visual) in the Neuropsychological Assessment Battery NAB

CONTACTS AND LOCATIONS:
Overall Officials: Grigore C Burdea, Ph.D., Study Chair — BRIGHT CLOUD INTL CORP
Locations (1):
- PowerBack Rehabilitation, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burdea G, Kim N, Polistico K, Kadaru A, Grampurohit N, Hundal J, Pollack S. Robotic Table and Serious Games for Integrative Rehabilitation in the Early Poststroke Phase: Two Case Reports. JMIR Rehabil Assist Technol. 2022 Apr 13;9(2):e26990. doi: 10.2196/26990. PMID 35416787
- See also: BCI's corporate site — http://www.BrightBrainer.com

DOCUMENTS (2):
  • Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04252170/ICF_000.pdf
  • Study Protocol (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/70/NCT04252170/Prot_001.pdf